CLINICAL TRIAL: NCT02398461
Title: A Double-Blind, Placebo-Controlled, Single Ascending Dose Intravenous Infusion Study of rHIgM22 in Patients With Multiple Sclerosis Immediately Following a Relapse
Brief Title: An Intravenous Infusion Study of rHIgM22 in Patients With Multiple Sclerosis Immediately Following a Relapse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM22-MS-1033
Record Dates: First submitted 2015-03-13; First posted 2015-03-25 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis, Acute Relapsing
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rHIgM22 (Experimental): Patients will be enrolled sequentially in 2 separate cohorts, representing escalating dose levels. Each dose cohort will comprise 15 subjects, randomly assigned to receive either rHIgM22 (n=10) or placebo (n=5).
  Interventions: Drug: rHIgM22
- Placebo (Placebo Comparator): Patients will be enrolled sequentially in 2 separate cohorts, representing escalating dose levels. Each dose cohort will comprise 15 subjects, randomly assigned to receive either rHIgM22 (n=10) or placebo (n=5).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rHIgM22 — Administered via IV infusion
  Other Names: M22
  Arms: rHIgM22
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, multi-center, double-blind, randomized, placebo-controlled, dose-escalation study in subjects with relapsing Multiple Sclerosis (MS). The primary outcome will be the safety and tolerability of a single dose of rHIgM22 in relapsing MS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (18-70 years of age; < 104 kg)
* Capable of giving informed consent
* Meet diagnostic criteria for MS, as defined by revised (2010) McDonald criteria
* Present with a clinical acute relapse defined as a new or worsening neurological symptoms attributable to MS preceded by a stable or improving neurological state of at least 30 days, not associated with fever or infection, lasting at least 24 hours and accompanied by an objective physical (neurological) exam finding as confirmed by the Investigator
* Has at least one new, identifiable, measurable and active lesion on MRI (Gd+) meeting the criteria of the imaging charter.

Exclusion Criteria:

* Certain specified co-morbidities (including pregnancy)
* Taking certain proscribed medications
* A medical regimen that has changed in the month prior to screening
* Inability to undergo requisite MRI evaluations
* Drug or alcohol abuse
* Any other reason for which, in the opinion of the Investigator, the subject should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses of rHIgM22 in patients with MS immediately following a relapse as measured by the number of patients with Adverse Events (AEs) | Up to 180 days
  Assessed by review of the AEs, including Serious Adverse Events (SAEs), clinical symptoms and signs, clinical laboratory tests and Electrocardiogram (ECGs).

SECONDARY OUTCOMES:
Maximum measured plasma concentration (Cmax) of single ascending doses of rHIgM22 | Pre-dose (day 1), specified time points up to 48 hours post treatment
Time to maximum plasma concentration (Tmax) of single ascending doses of rHIgM22 | Pre-dose (day 1), specified time points up to 48 hours post treatment
Half-life (T1/2) of single ascending doses of rHIgM22 | Pre-dose (day 1), specified time points up to 48 hours post treatment
Area under the concentration curve from time 0 to the concentration at last time point (AUC0-last) of single ascending doses of rHIgM22 | Pre-dose (day 1), specified time points up to 48 hours post treatment
Immunogenicity profile of single ascending doses of rHIgM22 | Specified time points up to 180 days post treatment
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies.
The Expanded Disability Status Scale (EDSS) | Screening, specified time points up to 180 days post treatment

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Acorda Site #12, Long Beach, California
  - Acorda Site #3, Sacramento, California
  - Acorda Site #7, San Francisco, California
  - Acorda Site #11, Aurora, Colorado
  - Acorda Site #16, Centennial, Colorado
  - Acorda Site #22, Chicago, Illinois
  - Acorda Site #14, St Louis, Missouri
  - Acorda Site #19, Teaneck, New Jersey
  - Acorda Site #10, Rochester, New York
  - Acorda Site #18, Dallas, Texas
  - Acorda Site #2, Seattle, Washington
  - Acorda Site #6, Seattle, Washington

REFERENCES:
- [Derived] Greenberg BM, Bowen JD, Alvarez E, Rodriguez M, Caggiano AO, Warrington AE, Zhao P, Eisen A. A double-blind, placebo-controlled, single-ascending-dose intravenous infusion study of rHIgM22 in subjects with multiple sclerosis immediately following a relapse. Mult Scler J Exp Transl Clin. 2022 Apr 26;8(2):20552173221091475. doi: 10.1177/20552173221091475. eCollection 2022 Apr-Jun. PMID 35496758